CLINICAL TRIAL: NCT06161805
Title: Esketamine as Treatment for Chronic Pain Due to Endometriosis: a RCT Study
Acronym: EASYlight
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Reinier de Graaf Groep (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EASYlight-NEK
Record Dates: First submitted 2023-10-23; First posted 2023-12-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis; Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Endometriosis | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Care Provider, Investigator
Masking Description: The researchers and participants will not be informed on the nature of the treatment until the trial is fully completed, and the database is locked. Only the clinical pharmacist who prepares the study medication will be aware of the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine (Experimental): Esketamine dosing regimen is set at 0.1 mg/kg/h as starting dosage. Dosage will be gradually increased based on heart rate, oxygen saturation, blood pressure and side effects (e.g. nausea and dissociative effects) during a period of 8 hours to a maximum of 0.5 mg/kg/h (in steps of 0.1-0.3-0.5 mg/kg/hour).
  Interventions: Drug: Esketamine hydrochloride
- Placebo (Placebo Comparator): 8 hours infusion with saline (NaCl 0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esketamine hydrochloride — Esketamine dosing regimen is set at 0.1 mg/kg/h as starting dosage. Dosage will be gradually increased based on heart rate, oxygen saturation, blood pressure and side effects (e.g. nausea and dissociative effects) during a period of 8 hours to a maximum of 0.5 mg/kg/h (in steps of 0.1-0.3-0.5 mg/kg/hour). This dosage regimen is similar to that used earlier by Sigtermans et al. [1].
  Other Names: ketanest
  Arms: Esketamine
Drug: Placebo — 8 hour infusion with saline (NaCl 0.9%)
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled trial is to investigate the effect of esketamine versus placebo on the NRS score for chronic pelvic pain. Secondary endpoints are to assess pain scores, side-effects, quality of life, depressive symptoms and pain coping.

DETAILED DESCRIPTION:
Endometriosis is a chronic inflammatory disease affecting approximately 10% of reproductive-aged women. Severe pain symptoms and subfertility result in a lower quality of life, higher prevalence of depression and loss of productivity. Consequently, the economic impact of endometriosis is high. Treatment options to suppress chronic pain symptoms in patients with (deep) endometriosis are inadequate, resulting in increased opioid consumption. Ketamine (in our study we will use the S-enantiomer, esketamine), is a versatile drug with analgesic, anti-inflammatory and antidepressant effects and is commonly used in the treatment of chronic pain patients and has shown promising outcomes. However, whilst esketamine targets multiple aspects of endometriosis simultaneously (pain, inflammation, depression), studies on esketamine as treatment for chronic pain due to endometriosis have never been reported. Therefore we aim to conduct a randomized controlled trial to assess the efficacy of esketamine infusion versus placebo in the treatment of chronic endometriosis-induced pain.

ELIGIBILITY:
Inclusion Criteria:

* Women
* All pre-menopausal women aged above 18 years
* Diagnosed with endometriosis (ultrasound, MRI or previous laparoscopic and/or diagnostic surgery) according to the #Enzian classification [52]. This means that endometriosis is present in the following compartments:

  * Rectovaginal space (minimal A1) and/or
  * Sacrouterine ligaments, cardinal ligaments, pelvic sidewall (minimal B1) and/or
  * Rectum (minimal C1) and/or
  * Endometriosis of the intestines, diaphragm and/or
  * Adenomyosis (according to the morphological uterus sonographic assessment (MUSA) or evident adenomyosis on the MRI) [53, 54] and/or
  * Peritoneal / superficial endometriosis (diagnosed laparoscopically and not treated during surgery).
* Mild to severe chronic pelvic pain (NRS scale >= 6). The 11-point NRS scale ranges from '0' representing no pain to '10' representing the worst pain imaginable.
* Resistant to current recommended lines of analgesics (paracetamol, NSAIDs)
* Usage of strong opioids must not have been prescribed or otherwise have been discontinued for more than 1 week.
* An indication for endometriosis resection surgery or on the waiting list for surgical treatment
* Ability to understand the patient information letter and to give oral and written informed consent
* No alteration in the utilization of hormonal therapy ≤1 months prior to inclusion.

Exclusion Criteria:

* Pain score <6 out of 10 (NRS) for chronic pelvic pain
* Endometriosis affecting the bladder and ureter
* Increased intracranial pressure
* Poorly regulated hypertension, >180/100mmHg at rest
* Patients with thyroid disease
* Patients with cancer
* History of psychiatric illness (schizophrenia, psychosis, delirium, manic depression)
* Serious medical disease (e.g., cardiovascular, renal , pulmonary or liver disease)
* Severe liver disease
* Patients with glaucoma
* Usage of strong opioid medication
* Usage of xanthine derivatives or ergometrine
* Unstable angina, heart failure, history of cerebral vascular accident (CVA)
* Patients suffering from an active infection
* Patients with epilepsy
* Patients trying to achieve pregnancy and or patients who are breastfeeding
* Not being able to answer questionnaires (in Dutch)
* Mentally incompetent (patients not able to make decisions that are in their best interests, this will be evaluated by their treating physician (e.g. patients with an intellectual disability or mental retardation))
* Alcohol or drug abuse
* Patient with a known (es)ketamine allergy
* Abnormal liver enzyme levels at baseline (ASAT, ALAT, GGT, AF, Bilirubin total)

Patients are allowed to continue the following pain medications: paracetamol, non-steroidal anti-inflammatory drugs as described previously by Sigtermans et al. (Trial NL466 (NTR507))* according to their stable use in dose and frequency.

*in case of tramadol, amitriptylin, selective serotonin reuptake-inhibitors, gabapentin and pregabalin, the usage may also be continued during this study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Endometriosis is a condition exclusive to females
Enrollment: 56 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Chronic pelvic pain | 4 weeks after the 8 hour infusion treatment.
  The effect of treatment allocation on the NRS score for chronic pelvic pain. The NRS scale ranges from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Dysmenorrhea | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  NRS score for dysmenorrhea. The NRS scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Dyschezia | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  NRS scores for dyschezia.The NRS scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Dysuria | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  NRS scores for dysuria. The NRS scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Dyspareunia | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  NRS score for dyspareunia. The NRS scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Chronic pelvic pain | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  NRS score for chronic pelvic pain. The NRS scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Depressive symptoms | Baseline, 4 weeks after infusion treatment
  Hospital Anxiety and Depression scale, 14 questions, scale from 0-3, higher scores mean worse outcome.
Endometriosis associated Quality of Life | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  Endometriosis Health Profile-30 (EHP-30). The overall EHP-30 score ranges from 0 to 100, with a high score indicating poorer health-related quality of life.
Quality of life in general | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  EuroQql five-dimensional 5 levels (EQ-5D-5L). According to the Dutch scoring algorithm, the EQ-5D-5L score index value ranges from -0.446 (55555 worst health state) to 1 (11111, best health state).
Quality of life in general | Baseline and week 4, 8, 12 after the 8 hour infusion treatment
  EuroQql Visual Analog Scale (EQ-VAS). Overall health will be represented by the EQ-VAS, ranging from 0 to 100, with higher scores indicating better health.
Productivity costs | 12 weeks post-infusion treatment
  Adjusted productivity costs questionnaire (iPCQ): institute for Medical Technology Assessment (iMTA). Adjusted medical consumption questionnaire: iMTA. Productivity costs will be measured by calculating absence from paid work (absenteeism), reduced productivity at paid work (presenteeism), and productivity loss in unpaid work. Hours of productivity loss will be translated by a standard cost price of productivity per hour.
Medical costs | Baseline, 12 weeks post-infusion treatment
  Medical consumption costs will be calculated based upon the iMCQ.
Pain coping and cognition | Baseline, 12 weeks post-infusion treatment
  Pain Coping and Cognition list (PCCL), consists of 42 items divided in four scales: pain catastrophising (higher scores mean a higher degree of catastrophising), pain coping (lower scores mean a lower degree of pain coping), internal pain control (lower scores mean less internal pain control) and external pain control (higher scores mean less external pain control.
The effect infusion treatment psychedelic effects | On the day of infusion (prior to infusion and during infusion)
  Bowdle questionnaire, scale from 0-100, higher scores mean worse outcome.
Treatment experience | Directly after infusion
  1 question, treatment rating on a scale from 0 (worst experience possible) -10 (excellent experience)

CONTACTS AND LOCATIONS:
Locations (1):
- Nederlandse Endometriose Kliniek, Reinier de Graaf Gasthuis, Delft, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
upon request

REFERENCES:
- [Background] Sigtermans MJ, van Hilten JJ, Bauer MCR, Arbous SM, Marinus J, Sarton EY, Dahan A. Ketamine produces effective and long-term pain relief in patients with Complex Regional Pain Syndrome Type 1. Pain. 2009 Oct;145(3):304-311. doi: 10.1016/j.pain.2009.06.023. Epub 2009 Jul 14. PMID 19604642